CLINICAL TRIAL: NCT02487563
Title: A Prospective Study of Patients With Isolated Thrombocytopenia Following Hematopoietic Stem Cell Transplantation
Brief Title: Prospective Study of Patients With Thrombocytopenia Following HSCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Peking University People's Hospital (Other); Nanfang Hospital, Southern Medical University (Other); Ruijin Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Qilu Hospital of Shandong University (Other); Children's Hospital of Soochow University (Other); Fujian Medical University Union Hospital (Other); Hebei Yanda Ludaopei Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOOCHOW-HY-2015
Record Dates: First submitted 2015-06-21; First posted 2015-07-01 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-04

CONDITIONS: Thrombocytopenia; Hematologic Diseases
Keywords: Isolated thrombocytopenia; decitabine; rhTPO
MeSH Terms: conditions — Thrombocytopenia; Hematologic Diseases | interventions — Decitabine; Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Experimental Group 1 (Experimental): Decitabine in combination with rhTPO.
  Interventions: Drug: Decitabine; Drug: rhTPO
- Experimental Group 2 (Experimental): Decitabine
  Interventions: Drug: Decitabine
- Control Group (Active Comparator): Conventional treatment except decitabine.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Drug: Decitabine — Decitabine
  Other Names: 5-Aza-2'-deoxycytidine
  Arms: Experimental Group 1; Experimental Group 2
Drug: rhTPO — rhTPO
  Other Names: Thrombopoietin
  Arms: Experimental Group 1
Other: Conventional Treatment — immunoglobulin, glucocorticoid etc
  Arms: Control Group

SUMMARY:
Isolated thrombocytopenia is a common and severe complication of HSCT, which often leads to an increased risk of life-threatening hemorrhage, frequent requirement of platelet transfusions and extended hospital stays, representing a challenging clinical problem. Current treatments for thrombocytopenia after HSCT are frequently unsatisfactory in platelet recovery and for preventing potentially fatal bleeding complications. Therefore, it is urgent to explore an effective therapy to improve the outcomes of thrombocytopenia after HSCT. Previous studies have demonstrated that decitabine, a hypomethylating agent, may reduce platelet transfusions in myelodysplastic syndrome (MDS) patients. The investigators conducted an prospective clinical trial to evaluate the safety and efficiency of rhTPO and decitabine in the treatment of thrombocytopenia following HSCT.

DETAILED DESCRIPTION:
Isolated thrombocytopenia is a frequent and severe complication of hematopoietic stem cell transplantation (HSCT). It often leads to an increased risk of life-threatening hemorrhage, frequent requirement of platelet transfusions and extended hospital stays, representing a challenging clinical problem. Current treatments for thrombocytopenia after HSCT, including thrombopoietin, interleukin-11, immunoglobulin, methylprednisolone and rituximab, are frequently unsatisfactory in platelet recovery. Therefore, it is urgent to explore an effective therapy to improve the outcomes of thrombocytopenia after HSCT. Thrombopoietin (TPO) is a cytokine that drives thrombopoiesis by stimulating the differentiation of stem cells into megakaryocytes and promoting megakaryocyte proliferation and polyploidization. Decitabine was approved for the treatment of myelodysplastic syndrome (MDS) as a DNA methylation inhibitors. Studies in vitro show that decitabine enhances platelet release and megakaryocyte maturation. Here, the investigators performed a prospective clinical trial, in order to investigate the safety and efficiency of rhTPO and decitabine in the treatment of thrombocytopenia following HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Platelet count ≤ 30 × 109/L persistently at day 60 post-HSCT or later;
2. Neutrophil and hemoglobin were well recovered;
3. Full donor chimerism was achieved;
4. No response to conventional treatments (e.g. thrombopoietin, immunoglobulin, glucocorticoid alone or in combination) for a duration of at least 4 weeks;

Exclusion Criteria:

1. Patients with malignancy relapse;
2. Active infections;
3. Grade Ⅲ-Ⅳ acute GVHD or severe chronic GVHD according to National Institute of Health criteria;
4. Severe organ damage;
5. Thrombosis requiring treatment;
6. Received decitabine following the current transplantation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2015-10; Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Depei Wu, PhD,MD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First affiliated Hospital of SooChow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] First LR, Smith BR, Lipton J, Nathan DG, Parkman R, Rappeport JM. Isolated thrombocytopenia after allogeneic bone marrow transplantation: existence of transient and chronic thrombocytopenic syndromes. Blood. 1985 Feb;65(2):368-74. PMID 3881142
- [Result] Wang J, Yi Z, Wang S, Li Z. The effect of decitabine on megakaryocyte maturation and platelet release. Thromb Haemost. 2011 Aug;106(2):337-43. doi: 10.1160/TH10-11-0744. Epub 2011 Jun 28. PMID 21713321
- [Result] Zhou H, Hou Y, Liu X, Qiu J, Feng Q, Wang Y, Zhang X, Min Y, Shao L, Liu X, Li G, Li L, Yang L, Xu S, Ni H, Peng J, Hou M. Low-dose decitabine promotes megakaryocyte maturation and platelet production in healthy controls and immune thrombocytopenia. Thromb Haemost. 2015 May;113(5):1021-34. doi: 10.1160/TH14-04-0342. Epub 2015 Jan 8. PMID 25566808
- [Derived] Tang Y, Chen J, Liu Q, Chu T, Pan T, Liang J, He XF, Chen F, Yang T, Ma X, Wu X, Hu S, Cao X, Hu X, Hu J, Liu Y, Qi J, Shen Y, Ruan C, Han Y, Wu D. Low-dose decitabine for refractory prolonged isolated thrombocytopenia after HCT: a randomized multicenter trial. Blood Adv. 2021 Mar 9;5(5):1250-1258. doi: 10.1182/bloodadvances.2020002790. PMID 33646303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two participants from different institutions submitted the applications at the same time when there was only one quota left. Both of them met the inclusion criteria and were enrolled.
Period: Overall Study
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Started | 32 | 33 | 32
Completed | 30 | 30 | 31
Not Completed | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group 1: Decitabine 15 mg/m2 daily intravenously for consecutive 3 days (day 1 to day 3), combined with rhTPO 15000 U daily subcutaneously beginning on day 4 and continuing until the response was achieved or the time of initial evaluation.
- Experimental Group 2: Decitabine 15 mg/m2 daily intravenously for consecutive 3 days (day 1 to day 3) alone.
- Control Group: Conventional therapies with recommended options including rhTPO, eltrombopag, immunoglobulin, rituximab, interleukin-11 and glucocorticoids, alone or in combination.
- Total: Total of all reporting groups
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [23 to 43] | 36 [27 to 46] | 36 [28 to 51] | 31 [25 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 15 | 32
  Male | 25 | 18 | 16 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 30 | 30 | 31 | 91
Diagnosis [Count of Participants; unit: Participants]
  Acute lymphocytic leukemia | 8 | 10 | 11 | 29
  Acute myeloid leukemia | 15 | 14 | 12 | 41
  Chronic myeloid leukemia | 0 | 2 | 1 | 3
  Myelodyplastic syndrome | 5 | 4 | 4 | 13
  Non-Hodgkin lymphoma | 2 | 0 | 3 | 5
Transplant Donor [Count of Participants; unit: Participants]
  Haploidentical donor | 23 | 20 | 21 | 64
  Matched related donor | 5 | 8 | 6 | 19
  Matched unrelated donor | 2 | 2 | 4 | 8
ABO compatitibilty [Count of Participants; unit: Participants]
  ABO matched | 15 | 13 | 18 | 46
  ABO mismatched | 15 | 17 | 13 | 45
Conditioning [Count of Participants; unit: Participants]
  Busulfan / cyclophosphamide | 26 | 27 | 29 | 82
  Others | 4 | 3 | 2 | 9
Mononuclear cell infused [Median (Inter-Quartile Range); unit: 10E8/kg] | 9.78 [6.18 to 11.52] | 10.50 [7.77 to 12.55] | 9.40 [6.46 to 11.40] | 10.04 [6.82 to 12.29]
Neutrophils recovery [Median (Inter-Quartile Range); unit: days] | 12 [11 to 13] | 12 [12 to 14] | 13 [12 to 14] | 12 [12 to 14]
Enrollment time [Median (Inter-Quartile Range); unit: days] | 103 [71 to 149] | 105 [78 to 184] | 79 [63 to 129] | 99 [66 to 158]
Platelet counts at enrollment [Median (Inter-Quartile Range); unit: 10E9 platelets/L] | 14 [11 to 17] | 12 [9 to 17] | 17 [9 to 22] | 15 [10 to 18]
Megakaryocyte counts at enrollment [Median (Inter-Quartile Range); unit: cells/cm^2] | 2.9 [1.3 to 5.4] | 3.2 [1.8 to 6.1] | 3.1 [1.7 to 6.4] | 3.0 [1.5 to 6.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Platelet Count Recovery
Description: Platelet response refers to a sustained increase (stable or increasing level) of at least 30×10E9/L independent of transfusion for 3 days.
Time Frame: Up to 4 weeks after the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 30 | 30 | 31
Participants | 20 | 22 | 6

2. Secondary Outcome: Megakaryocyte Count
Description: The total number of megakaryocytes as well as the platelet-shedding megakaryocytes of bone marrow smears (per cm2) was counted and cross-checked by blinded observers.
Time Frame: Up to 4 weeks after the treatment
Measure: Median (Inter-Quartile Range); unit: cells/cm^2
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
Number analyzed (Participants) | 30 | 30 | 31
cells/cm^2 | 6.7 [1.2 to 10.0] | 7.5 [3.1 to 14.1] | 3.3 [1.8 to 6.0]

ADVERSE EVENTS:
Time Frame: Study period (4 weeks)
Arm/Group | Experimental Group 1 | Experimental Group 2 | Control Group
All-Cause Mortality (participants affected / at risk) | 1/30 | 0/30 | 1/31
Serious Adverse Events (participants affected / at risk) | 4/30 | 1/30 | 3/31
Other Adverse Events (participants affected / at risk) | 8/30 | 5/30 | 7/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group 1 (N=30) | Experimental Group 2 (N=30) | Control Group (N=31)
Bleeding events (Blood and lymphatic system disorders) | 1 | 1 | 0 — Bleeding events (grade ≥3)
Infections (Infections and infestations) | 2 | 0 | 2 — Infections (Grade >=3)
Shock (Cardiac disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group 1 (N=30) | Experimental Group 2 (N=30) | Control Group (N=31)
Hypohepatia (Hepatobiliary disorders) | 2 | 1 | 1
Chest distress (Cardiac disorders) | 1 | 1 | 0
Anorexia (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Fever (Infections and infestations) | 1 | 2 | 1
Blurred vision (Eye disorders) | 0 | 1 | 0
Hypeluricemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Erythra (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Bleeding events (Blood and lymphatic system disorders) | 3 | 2 | 3
Infection (Infections and infestations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Small number of patients, the diversity of patients, and the heterogeneous treatment options in Arm C.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02487563/Prot_SAP_ICF_000.pdf